CLINICAL TRIAL: NCT05023057
Title: A Multicenter Randomized Controlled Study to Evaluate the Efficacy of a 24-week Multidomain Intervention Via Face-to-face and Video Communication Platforms in Mild Cognitive Impairment
Brief Title: Multidomain Interventions Via Face-to-face and Video Communication Platforms in Mild Cognitive Impairment
Acronym: SUPERBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Seong Hye Choi, MD, Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-06-040
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: outcome assessor-blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidomain intervention (Experimental): The participants in the intervention arm will receive all five components of the intervention: (1) monitoring and management of metabolic and vascular risk factors; (2) cognitive training and social activity; (3) physical exercise; (4) nutritional guidance; and (5) motivational training.
  Interventions: Behavioral: Multidomain intervention
- Control (No Intervention): At baseline, the participants in the control group will meet a study doctor, be prescribed medication when necessary, and receive educational booklets corresponding to their risk factors and a booklet on lifestyle guidelines to prevent dementia. They will receive usual care during the study period and be informed that they could participate in the multidomain intervention program after this study end.

INTERVENTIONS:
Behavioral: Multidomain intervention — For 24 weeks, participants will receive cognitive training using the tablet PC application twice a week, exercise 3 times a week, nutrition education 12 times, anthropometric measurements and alcohol and smoking monitoring every 4 weeks, motivation reinforcement training 4 times.
  Arms: Multidomain intervention

SUMMARY:
This study will be done to investigate the effectiveness of a 24-week multidomain intervention program consisting of cognitive training, exercise, nutrition management, vascular disease risk factor management, social activity, and motivational enhancement on the cognitive function compared to the control group in mild cognitive impairment.

DETAILED DESCRIPTION:
The physical exercise program will consist of aerobic exercise, exercise to enhance balance and flexibility, muscle-strengthening activities involving major muscle groups, and finger-toe movements. Cognitive training targets the cognitive domains of episodic memory, executive function, attention, working memory, calculation, and visuospatial function. Cognitive training will be conducted using a tablet-based application. Participants will be advised to eat something according to the recommendation of the MIND diet. They will also meet the study nurse every 4 weeks for anthropometric measurements and monitoring of smoking and alcohol intake. The purpose of the motivational enhancement program is to induce, maintain, and strengthen motivation, which is a psychological resource to help maintain dementia prevention activities.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 85 years of age
* Having at least one modifiable dementia risk factor
* Complaints of cognitive decline by a participant or informant
* A performance score that is lower than 1.0 standard deviations below the age-, and education-adjusted normative means for one or more of the delayed recall, naming, visuoconstruction, attention, and executive function tests
* MMSE Z score ≥ - 1.5
* Independent activities of daily living
* Being able to use the tablet PC through education, or having a person who can help a participant use the tablet PC.
* Having a reliable informant who could provide investigators with the requested information
* Provide written informed consent

Exclusion Criteria:

* Major psychiatric illness such as major depressive disorders
* Dementia
* Other neurodegenerative disease (e.g., Parkinson's disease)
* Malignancy within 5 years
* Cardiac stent or revascularization within 1 year
* Serious or unstable symptomatic cardiovascular disease
* Other serious or unstable medical disease such as acute or severe asthma, active gastric ulcer, severe liver disease, or severe renal disease
* Severe loss of vision, hearing, or communicative disability
* Any conditions preventing cooperation as judged by the study physician
* Significant laboratory abnormality that may result in cognitive impairment
* Illiteracy
* Unable to participate in exercise program safely
* Coincident participation in any other intervention trial

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change of cognition | Change from Baseline at 24 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status (range 40-160). Higher scores indicate better performance.

SECONDARY OUTCOMES:
Change of global cognition | Change from Baseline at 24 weeks
  Mini-Mental State Examination (range 0-30). Higher scores indicate better performance.
Change of function | Change from Baseline at 24 weeks
  Clinical Dementia Rating scale-Sum of Boxes (range 0-18). Higher scores indicate worse performance.
Change of subjective memory | Change from Baseline at 24 weeks
  Prospective and Retrospective Memory Questionnaire (range 16-80). Higher scores indicate worse performance.
Change of depression | Change from Baseline at 24 weeks
  Geriatric Depression Scale-15 items (range 0-15). Higher scores indicate worse performance.
Change of quality of life | Change from Baseline at 24 weeks
  Quality of life-Alzheimer's disease (range 0-52). Higher scores indicate better performance.
Change of activities of daily living | Change from Baseline at 24 weeks
  Bayer Activities of Daily Living (range 1-10). Higher scores indicate worse performance.
Change of nutritional behavior | Change from Baseline at 24 weeks
  Nutrition Quotient for elderly (range 0-100). Higher scores indicate better performance.
Change of nutrition | Change from Baseline at 24 weeks
  Mini Nutritional Assessment (range 0-14). Higher scores indicate better performance.
Change of motor function | Change from Baseline at 24 weeks
  Short Physical Performance Battery (range 0-12). Higher scores indicate better performance.
Change of sleep quality | Change from Baseline at 24 weeks
  Pittsburgh Sleep Quality Index (range 0-21). Higher scores indicate worse performance.
Change of motivation | Change from Baseline at 24 weeks. Higher scores indicate better performance.
  Self Determination Index (SDI). Higher scores of SDI indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hye Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (17):
- South Korea (17):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Myungji Hospital, Goyang-si
  - Chonnam University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Catholic Kwandong University International St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Bobath Memorial Hospital, Seongnam
  - CHA Bundang Medical Center, Seongnam
  - Ewha Womans Seoul Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 2 years since March 2024.
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Hwang J, Moon SY, Lee H, Lee J, Park YK, Jeong JH, Hong CH, Jung J, Na HR, Cho SH, Sung J, Lee SJ, Choi SH. Polygenicity and APOE epsilon4 shape response to intervention in mild cognitive impairment. Alzheimers Res Ther. 2025 Dec 12;17(1):262. doi: 10.1186/s13195-025-01907-3. PMID 41388319
- [Derived] Moon SY, Park YK, Jeong JH, Hong CH, Jung J, Na HR, Cho SH, Kim HS, Song HS, Choi M, Ku BD, Moon YS, Han HJ, Hong YJ, Kim EJ, Kim GH, Kim KW, Jang H, Yoon SJ, Kim HJ, Choi SH. South Korean study to prevent cognitive impairment and protect brain health through multidomain interventions via face-to-face and video communication platforms in mild cognitive impairment (SUPERBRAIN-MEET): A randomized controlled trial. Alzheimers Dement. 2025 Feb;21(2):e14517. doi: 10.1002/alz.14517. Epub 2025 Jan 22. PMID 39840755
- [Derived] Cho SH, Kang HJ, Park YK, Moon SY, Hong CH, Na HR, Song HS, Choi M, Jeong S, Park KW, Kim HS, Chun BO, Jung J, Jeong JH, Choi SH. SoUth Korean study to PrEvent cognitive impaiRment and protect BRAIN health through Multidomain interventions via facE-to-facE and video communication plaTforms in mild cognitive impairment (SUPERBRAIN-MEET): Protocol for a Multicenter Randomized Controlled Trial. Dement Neurocogn Disord. 2024 Jan;23(1):30-43. doi: 10.12779/dnd.2024.23.1.30. Epub 2024 Jan 29. PMID 38362052